CLINICAL TRIAL: NCT04884438
Title: A Brief Intervention for the Promotion of Wellbeing: the Power of Gratitude
Brief Title: Intervention for the Promotion of Gratitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gratitude
Record Dates: First submitted 2021-05-05; First posted 2021-05-13 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Affect
Keywords: Gratitude; Wellbeing; Positive affect; Ecological momentary assessment
MeSH Terms: interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Psychological intervention for the promotion of gratitude — A brief intervention protocol has been developed for the promotion of gratitude. The protocol is manualized and the content will be explained to each participant in the videoconference sessions, and a copy of the manual will be given (or sent) to the patients at the end of the therapy sessions.
  The structure and contents of the intervention are summarized below:
  1. Psychoeducation about gratitude and its effects on health (both physical and psychological).
  2. Gratitude towards life:
     1. Gratitude walk
     2. Three positive things
     3. Sharing gratitude
  3. Social gratitude:
     1. Daily thanks to others
     2. Gratitude letter
     3. Proof of gratitude
  4. Self-gratitude: this part includes an exercise aimed at fostering self-gratitude in three different areas:
     1. Gratitude for the things I do to take care of my physical health.
     2. Gratitude for what I do to take care of my mental health, my self-esteem and my personal development.
     3. Gratitude for what I do to take care of others.

SUMMARY:
This study aims to analyze the effects of a psychological intervention to promote wellbeing. To do so, a brief intervention is developed to enhance a sense of gratitude through a multiple baseline across components design. Traditional measures will be used together with the incorporation of a novel evaluation methodology such as the EMA, which allows the collection of data in the context of people's daily lives and at different specific times, that is, in real time.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* A score of, at least, 1 standard deviation below the mean for the PANAS positive subscale, based on the norms of the general population

Exclusion Criteria:

* Suicide risk
* Bipolar disorder
* Psychosis
* Any medical or psychiatric condition that hinders participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative Affect Schedule (PANAS) (Watson, Clark, & Tellegen, 1988; Spanish version: Sandín et al., 1999) at pre-intervention, during the intervention, post-intervention, and 1-month follow-up. | Up to 2 months
  The PANAS consists of 20 items with a range from 1 (very slightly or not at all) to 5 (extremely). Respondents have to indicate the extent to which they experienced the feeling or emotion during the past few weeks. This scale evaluates two independent dimensions: positive affect and negative affect. The maximum score for each subscale is 50. The scale showed excellent internal consistency (α between .84 and .90) and convergent and discriminant validity. The Spanish version has demonstrated high internal consistency (α = 0.89 and 0.91 for positive affect and negative affect in women, respectively, and α = 0.87 and 0.89 for PA and NA in men, respectively) in college students.
Change in Gratitude Questionnaire 6-item (GQ-6) (McCullough, Emmons, & Tsang, 2001; Spanish version: Magallares, Recio, & Sanjuán, 2018) at pre-intervention, during the intervention, post-intervention, and 1-month follow-up. | Up to 2 months
  The GQ-5 consists of six items that measure span, frequency, intensity and density of gratitude and primarily focuses on the unidimensional emotional component of gratitude. Participants have to rate six items (e.g., "I have so much in life to be thankful for") on a seven-point Likert scale (GQ-6: α = 0.82)

SECONDARY OUTCOMES:
Change in Satisfaction with life (SWLS) (Diener, Emmos, Larse, & Griffin, 1985; Spanish version: Vázquez, Duque, & Hervás, 2013) at pre-intervention, post-intervention, and 1-month follow-up. | Up to 2 months
  This is a life satisfaction scale consisting of five items. Participants are asked to indicate their degree of agreement with each statement using a 7-point Likert scale (from 1 = strongly disagree to 7 = strongly agree). Scores can range from 5 to 35 points, indicating a greater life satisfaction with higher scores (alpha = .88).
Change in Overall Anxiety Severity and Impairment Scale (OASIS) (Campbell-Sills et al., 2009; Spanish version: González-Robles et al., 2018) at at pre-intervention, during the intervention, post-intervention, and 1-month follow-up. | Up to 2 months
  The OASIS is a 5-item self-report scale that evaluates the frequency and severity of anxiety symptoms, the functional impairment related to these symptoms (i.e. school, work, home, or social impairment), and behavioral avoidance. Each item instructs respondents to endorse one of five responses that best describes their experiences over the past week. Response items are coded from 0 to 4, added together to obtain a total score ranging from 0 to 20. Previous studies have shown good internal consistency (α = 0.80), test-retest reliability, and convergent and discriminant validity. The Spanish version has shown good internal consistency (α = 0.86), and convergent and discriminant validity.
Change in Overall Depression Severity and Impairment Scale (ODSIS) (Bentley et al., 2014; Spanish version: Mira et al., 2019) at pre-intervention, during the intervention, post-intervention, and 1-month follow-up. | Up to 2 months
  The ODSIS is a brief self-reported scale with 5 items that assess the severity and functional impairment associated with depressive symptoms. Items are coded on a 5-point scale (0-4). The sum of the scores is used to obtain the total score, which can be a maximum of 20. The measure has shown excellent internal consistency (α = 0.94 in an outpatient sample, 0.92 in a community sample, and 0.91 in a student sample) and good convergent/discriminant validity. The Spanish validation has excellent internal consistency (α = 0.93), as well as convergent and discriminant validity.
Change in Pemberton Happiness Index (PHI) (Hervás & Vázquez, 2013) at pre-intervention, post-intervention, and 1-month follow-up. | Up to 2 months
  The Pemberton Happiness Index (PHI) is a self-reported scale of overall well-being that includes both remembered and experienced well-being. PHI index incorporates two components: (a) an 11-item measure that includes general, eudaimonic, hedonic, and social well-being rated on a scale from 0 to 10 (in this scale, participants are asked to rate each statement using a scale from 0 -fully disagree- to 10 -fully agree-) and (b) a single score that results from the combination of positive and negative experiences from the day before, also on a scale from 0 to 10. The scale has shown excellent internal consistency in Spanish samples (alpha between .91 and .92).
Change in Dispositional Hope Scale (DHS) (Snyder et al., 1991; Spanish version: Galiana et al., 2015) at pre-intervention, post-intervention, and 1-month follow-up. | Up to 2 months
  The Dispositional Hope Scale (DHS) is a 12-item instrument, with 4 pathways items, measuring abilities to identify feasible ways to goal, and four agency items, which evaluate motivations for pursuing goals, and four filler items. Items are scored in a scale from 1(definitely false) to 4 (definitely true). In the Spanish version, Cronbach's alphas ranged between .67 and .83.
Change in Subjective Happiness Scale (SHS) (Lyubomirsky & Lepper, 1999; Spanish version: Extremera & Fernández-Berrocal, 2014) at pre-intervention, post-intervention, and 1-month follow-up. | Up to 2 months
  The SHS is a 4-item Likert-type (from 1 to 7) scale measure that evaluates global subjective happiness using statements with which participants either self-rate themselves or compare themselves to others. The scale has an adequate unitary structure and temporal stability confirmed in 14 samples, showing moderate correlations with constructs such as self-esteem, depression, satisfaction, or neuroticism.
Change in Credibility/Expectancy Questionnaire (CEQ) (Devilly & Borkovec, 2000) at pre-intervention. | Baseline
  The scale comprises 6 items, rated on a scale from 0 (nothing at all) to 9 (completely), that cover how logical the treatment seems to be, how successfully the patients think the treatment will be in reducing their symptoms, how confident they are in recommending the treatment to a friend, how much improvement in their symptoms they think will occur, how much they really feel that therapy will help them to reduce their symptoms, and how much improvement in their symptoms they really feel will occur.

CONTACTS AND LOCATIONS:
Locations (1):
- Edificio de Investigación, Castellon, Spain

IPD SHARING:
Plan to Share IPD: No